CLINICAL TRIAL: NCT05001152
Title: An Open-Label Taste Assessment of Ozanimod in Healthy Subjects
Brief Title: Taste Assessment of Ozanimod
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM047-013
Record Dates: First submitted 2021-08-06; First posted 2021-08-11 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Healthy Volunteers
Keywords: Ozanimod
MeSH Terms: interventions — ozanimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ozanimod (Experimental): A maximum of 10 healthy adult participants (i.e., sensory panelists) will complete a maximum of 20 taste assessment days, with at least 4 panelists required to evaluate the taste characteristics of ozanimod on each taste assessment day.
  Interventions: Drug: Ozanimod

INTERVENTIONS:
Drug: Ozanimod — Taste assessment

SUMMARY:
The purpose of this study is to assess the taste characteristics of ozanimod formulations, alone and mixed, in order to develop a pediatric oral form of ozanimod.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, between 25 and 80 years of age.
* Participant is a qualified sensory panelist selected by Senopsys based on training and experience

Exclusion Criteria:

* Participant has any history of any illness, medical condition, laboratory abnormality, or psychiatric illness that might confound the results of the study or places the panelist at unacceptable risk if he or she were to participate in the study.
* Participant is a female that is pregnant, nursing, or planning to become pregnant during the study.

Other protocol-defined inclusion/exclusion criteria apply

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Taste evaluation - Aromatic identity | Up to 6 months
  Measured using the Flavor Profile method of descriptive sensory analysis
Taste evaluation - Amplitude | Up to 6 months
  Measured using the Flavor Profile method of descriptive sensory analysis
Taste evaluation - Off-notes | Up to 6 months
  Measured using the Flavor Profile method of descriptive sensory analysis
Taste evaluation - Aftertaste | Up to 6 months
  Measured using the Flavor Profile method of descriptive sensory analysis

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Local Institution - 0001, Woburn, Massachusetts
  - Senopsys LLC, Woburn, Massachusetts

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm